CLINICAL TRIAL: NCT04895111
Title: Role of Endobronchial Ultrasound Strain Elastography (EBUS-SE) in Sarcoidosis: a Prospective Cohort Study
Brief Title: Endobronchial Ultrasound Strain Elastography in Sarcoidosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 4066
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-08

CONDITIONS: Sarcoidosis, Pulmonary
Keywords: Sarcoidosis; Endobronchial Ultrasound; Elastography; Endosonography; Granuloma
MeSH Terms: conditions — Sarcoidosis, Pulmonary; Sarcoidosis; Granuloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with suspected sarcoidosis: Consecutive patients with clinical and radiological (CT scan +/- PET) suspect of sarcoidosis
  Interventions: Diagnostic Test: Endobronchial ultrasound strain elastography

INTERVENTIONS:
Diagnostic Test: Endobronchial ultrasound strain elastography — Measurement of tissue elasticity of hilar and mediastinal lymph nodes through strain elastography measured during an endonbronchial ultrasound examination

SUMMARY:
Strain elastography (SE) is an imaging method used for the measurement of relative tissue elasticity through qualitative (color pattern) or semi-quantitative methods (strain ratio or strain histogram). Very recently, the first pilot study has provided preliminary evidence that EBUS-SE elastography may help identify fibrotic lymph nodes in sarcoidosis and that sampling lymph nodes characterized by low strain elastography, that is "stiff" nodes, is associated with an increased risk of retrieving an inadequate sample (i.e. a sample which is not representative of the lymph node tissue). The investigators hypothesize that an EBUS-SE pattern indicative of lymph node stiffness will be associated with less granulomas and more fibrosis.

DETAILED DESCRIPTION:
In the last decade, the possibility to sample under ultrasound guidance (endosonography) the intrathoracic lymph nodes through the airways (endobronchial ultrasound guided, EBUS-TBNA) or through the oesophagus (endoscopic ultrasound-guided fine needle aspiration, EUS-FNA/EUS-b-FNA) has revolutionized the diagnostic approach to sarcoidosis. Individual studies and meta-analyses performed in selected and unselected patient populations have shown that EBUS and EUS both have overall diagnostic accuracy exceeding 80%. In addition, endosonography provides useful information about lymph node density; indeed, the presence of inhomogeneity in the lymph node texture on B-mode during endosonography represents the most important factor favouring infection over sarcoidosis in patients with lymphadenopathy.

Although the diagnostic success rate of EBUS-TBNA in detecting granulomas in lymph nodes of patients with suspected sarcoidosis is very high, the procedure is not foolproof and tends to have a lower yield in stages II/III as compared to stage I disease. Clinical experience suggests that at least some of the false-negative EBUS-TBNA results in sarcoidosis patients may be caused by the presence of lymph nodes with extensive fibrosis. We aim to evaluate whether EBUS-SE may help identify fibrotic lymph nodes in sarcoidosis and if the outcome of EBUS-TBNA is different in lymph nodes for which EBUS-SE suggest high fibrotic content.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* ASA physical status I-III.
* Clinical/radiological (computed tomography) suspicion of sarcoidosis (Stages I to III)

Exclusion Criteria:

* Inability or unwillingness to consent.
* Severe bleeding disorders
* Contraindication for temporary interruption of the use of anticoagulant or antiplatelet therapy different from aspirin.
* Recent and/or uncontrolled cardiac disease, uncontrolled pulmonary hypertension.
* Compromised upper airway (eg, concomitant head and neck cancer or central airway stenosis for any reason).
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a clinical and radiological suspect of sarcoidosis.
Sampling Method: Probability Sample
Enrollment: 701 (Estimated)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
• Diagnostic yield for the detection of granulomas on endosonography samples according to a mean value of the strain histogram <40 or ≥40 | 15 days
  The diagnostic yield for the detection of granulomas will be measured on a per lymph node basis (number of lymph nodes in which the pathological exam of endosonography samples identifies granulomas/number of lymph nodes submitted to endosonography)

SECONDARY OUTCOMES:
• Adequacy of endosonography samples according to a mean value of the strain histogram <40 or ≥40. | 15 days
  The adequacy will be measured on a per lymph node basis (number of lymph nodes in which the pathological exam shows an adequate endosonography sample/number of lymph nodes submitted to endosonography) and is defined as the presence of a preponderance of lymphocytes at the pathological exam of the endosonography sample.
• Correlation between the strain elastography pattern measured with the mean value of the strain histogram and the following variables: age, sex, sarcoidosis stage (I vs II vs III), duration of sarcoidosis-related symptoms. | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy